CLINICAL TRIAL: NCT05286034
Title: Artificial Intelligence-assisted Decision-making to Improve Women's Participation to Cervical Cancer Screening in Occitanie Region-France
Brief Title: Using Artificial Intelligence-based ChatBot to Improve Women's Participation to Cervical Cancer Screening Programme
Acronym: AppDate-You
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Centre Régional de Coordination des Dépistages des Cancers, centre-Carcassonne (Unknown); Université de Bretagne Occidentale, Brest-France (Unknown)
Responsible Party: Principal Investigator, Farida Selmouni, Principal Investigator, International Agency for Research on Cancer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IEC 21-16
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer Screening; Cervical Cancer
Keywords: cervical neoplasia; cervical cancer screening; chatbot; artificial intelligence; cluster randomized controlled trial; HPV vaginal self-sampling
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: A cluster randomized controlled trial with two arms (one experimental arm and one active control arm) will be conducted in the Occitanie region, France to assess the effectiveness of a decision aid accessible via artificial intelligence-based Chatbot platforms to improve the "return" rate of HPV self-samples and the proportion of invited women "well managed" among disadvantaged women. A cluster is defined by aggregated units for statistical information (Ilots Regroupés pour l'Information Statistique, IRIS) and it refers to a target size of 2000 inhabitants per unit. Only IRIS classified as 4 and 5 according to the French version of the European Deprivation Index (EDI) will be included. The study will be conducted as a two-armed nested into the French cervical cancer screening programme in the Occitanie Region. Clusters will be randomly assigned by a computer-generated randomized schedule following simple randomization procedures in a 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Women randomized to this group will be sent screening reminder letters to perform HPV self-sampling test, with access to a decision aid tool tailored to those with low education levels. This tool will be available via Chatbot platforms.
  Interventions: Behavioral: Decision aid tailored to women with lower educational attainment,accessible via artificial intelligence-based Chatbot platforms
- Control group (No Intervention): Women randomized to this group will be sent screening reminder letters to perform HPV self-sampling test (Standard care)

INTERVENTIONS:
Behavioral: Decision aid tailored to women with lower educational attainment,accessible via artificial intelligence-based Chatbot platforms — Non-compliant women those that have not been screened for more than 4 years and living in the disadvantaged areas will be sent screening reminder letters to perform HPV self-sampling (HPVss) test, with access to decision aid tailored to women with lower education attainment and available via Chatbot platforms.
  ChatBot will deliver information in a responsive, conversational way via text and spoken language in multiple languages through multiple mobile channels.
  Arms: Intervention group

SUMMARY:
This project looks to improve the return rate of HPV self-sampling (HPVss) as well as the management of women HPVss positive.

DETAILED DESCRIPTION:
France has already implemented a cervical screening programme based on HPV test for the whole female population aged 30-65 years. Non-participant women can perform HPV test at their home. However, less than 20% of French women performed vaginal self-sampling when a kit was sent to their home. Women with lower income and educational levels participate less to cervical screening. A variety of personal, practitioner, test-related and logistical barriers negatively impact the screening participation of French women. Key barriers to participation could be addressed by overcoming disparities in HPV-related knowledge and perceptions about cervical cancer screening. This study aims to evaluate the impact of sending HPV self-sampling kit at women's home, associated with providing, through multiple mobile channels, a multi-language decision aid designed for women with lower education accessible via artificial intelligence-based ChatBot. This decision aid will help women review high quality evidence on cervical cancer disease and screening modalities.

ELIGIBILITY:
Inclusion criteria: eligible women will be:

* aged 30-65
* did not perform a pap smear in the last 4 years
* are living in deprived clusters in the Occitanie region.
* did not answer to a first "invitation" letter to perform a clinician-collected HPV testing

Exclusion criteria: ineligible women will be those:

* outside the target age group
* had a Pap smear in the past 3 years
* had hysterectomy including cervix
* are pregnant
* already scheduled a screening appointment or had just attended a HPV screening
* had a cervical abnormality that was under exploration and/or treatment.
* participated to the study pilot

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3000 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
HPV self-sampling "return" rate | 1 year after postal mail
  Percent of women recalled who "return" HPVss over 12 months "Return" means: 1) the receipt of the vaginal self-sample at the laboratory; 2) the performance of clinician-collected HPV testing for those who prefer to be screened by a health professional; and 3) Information about a recent screening or a cervical screening exclusion reason.
Proportion of HPVss-positive women "well managed" | 1 year after postal mail
  Percent of recruited women well managed (Percent of women screened and completing full pathway of HPV screening and treatment over 12 months).
  "Well managed" is defined as: completed a valid screening test (sample processed successfully to positive or negative result, including recollection of invalid samples) AND
  * for HPV negative women, woman advised of negative result
  * for HPV positive women, completed assessment.
Cost and cost-efficacy | Month 36 - Month 48
  Costs will be estimated using an ingredients approach whereby resources used for the respective interventions are identified and valued. The incremental cost-effectiveness ratios (ICERs) will be calculated as the mean difference in total costs between the intervention groups with the mean difference in effects, and expressed as both euros and US dollars per percentage change in screening participation.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Régional de Coordination des Dépistages des Cancers-Centre d'Occitanie, Carcassone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Selmouni F, Guy M, Muwonge R, Nassiri A, Lucas E, Basu P, Sauvaget C. Effectiveness of Artificial Intelligence-Assisted Decision-making to Improve Vulnerable Women's Participation in Cervical Cancer Screening in France: Protocol for a Cluster Randomized Controlled Trial (AppDate-You). JMIR Res Protoc. 2022 Aug 2;11(8):e39288. doi: 10.2196/39288. PMID 35771872